CLINICAL TRIAL: NCT03361319
Title: A Phase I Trial of Combination Nab-Paclitaxel and Nintedanib or Nab-paclitaxel and Placebo in Relapsed Non-Small Cell Lung Cancer Adenocarcinoma
Brief Title: Combination Nab-paclitaxel (N-P) and Nintedanib or N-P and Placebo in Relapsed NSCLC Adenocarcinoma
Acronym: N3
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawal of financial support from funder
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Boehringer Ingelheim (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCR 4448
Record Dates: First submitted 2017-11-22; First posted 2017-12-04 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: NSCLC, Recurrent; Adenocarcinoma of Lung
Keywords: NSCLC; Non-Small Cell Lung Cancer; Adenocarcinoma of lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence; Adenocarcinoma of Lung | interventions — nintedanib; Albumin-Bound Paclitaxel; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Part I: A dose-escalation - standard 3+3 design. Part 2: A placebo-controlled, randomised, double-blind, 2-arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 2 only of the study is double-blinded. 2 arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: (Phase Ib) Dose Escalation (Experimental): A dose-finding study of nintedanib (Vargatef) with nab-paclitaxel (Abraxane) with a standard 3+3 design. In the dose escalation part there will be 3 dose cohorts of nintedanib:
  Dose level -1: 100mg po BID d2-7, 9-21, q21 Dose level 1: 150mg po BID d2-7, 9-21, q21 Dose level 2: 200mg po BID d2-7, 9-21, q21
  Interventions: Drug: Vargatef; Drug: Abraxane
- Part 1: Dose Expansion (Experimental): In the dose expansion part, 6 additional patients will be enrolled at the maximum tolerated dose (MTD) of nintedanib (Vargatef) with nab-paclitaxel (Abraxane), prior to proceeding to part 2.
  Interventions: Drug: Vargatef; Drug: Abraxane
- Part 2: (Phase II) (Placebo Comparator): A placebo-controlled, randomised, double-blind, 2-arm, phase 2 multi-centre clinical trial of nab-paclitaxel (Abraxane) with nintedanib (Vargatef) and nab-paclitaxel alone.
  Arm A: nab-paclitaxel + placebo Arm B: nab-paclitaxel + nintedanib
  Interventions: Drug: Vargatef; Drug: Abraxane; Other: placebo

INTERVENTIONS:
Drug: Vargatef — small molecule triple kinase inhibitor
  Other Names: Nintedanib; L01xe31
Drug: Abraxane — Paclitaxel formulated as albumin bound nanoparticles
  Other Names: Paclitaxel; L01CD01
Other: placebo — Placebo in place of Ninedanib
  Arms: Part 2: (Phase II)

SUMMARY:
A PHASE I/II TRIAL OF COMBINATION NAB-PACLITAXEL AND NINTEDANIB OR NAB-PACLITAXEL AND PLACEBO IN RELAPSED NSCLC ADENOCARCINOMA

DETAILED DESCRIPTION:
The study is divided into 2 parts: Part 1 is the Phase Ib portion of the trial and Part 2 is the Phase II portion of the trial. Once the Trial Steering Committee has completed the dose limiting toxicity (DLT) assessment for Part 1 and confirmed RP2D for Part 2, Part 2 enrolment will proceed. The objective(s) for each part are as follows:

Part 1: The objective of Part 1 is to evaluate the safety and tolerability of combination nab-paclitaxel and nintedanib in patients with stage IIIb and IV adenocarcinoma of the lung in second and third treatment line setting and to determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of nintedanib when given with nab-paclitaxel at 100mg/m2 d1, d8 q21.

Part 2: The primary objective of Part 2 is to explore the efficacy of combination nab-paclitaxel and nintedanib versus nab-paclitaxel and placebo in the same patient population, with nintedanib/placebo given at the recommended phase 2 dose (RP2D) as defined during part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 or over.
* Patients with a pathologically confirmed diagnosis of stage IIIb or stage IV adenocarcinoma of the lung; patients with locally recurrent disease (stage IIIa) and no radical treatment options are also eligible.
* Patients who have previously received no more than 2 lines of systemic therapy for NSCLC with palliative intent:
* Chemotherapy as first or second line with palliative intent
* Relapsing within 6 months of adjuvant chemotherapy after surgery or as part of radical chemo-radiotherapy, which count as one line of therapy
* Licenced or experimental maintenance therapy is allowed (e.g. pemetrexed)
* Immunotherapy at prior line of treatment (first or second line) is allowed.
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients with estimated life expectancy of ≥ 12 weeks.
* Patients with at least one radiologically measurable tumour lesion as defined by RECIST 1.1 criteria.
* Patients with adequate haematopoietic, hepatic and renal function.
* Signed informed consent in accordance with local legislation.

Exclusion Criteria:

* Patients with a known EGFR kinase sensitising mutation or ALK gene fusion prior to enrolment who have not received prior TKI (patients enrolled and subsequently found to be positive will remain on protocol). Patients with known EGFR activating mutation or ALK fusion who have received appropriate TKI treatment will be allowed.
* Any concurrent anticancer systemic therapy.
* Prior treatment with nintedanib or any other VEGFR inhibitor; prior treatment with bevacizumab is allowed
* Patients refractory to prior taxane therapy for advanced disease. Prior taxane used in the adjuvant setting does not exclude eligibility provided there is no disease recurrence within 12 months upon completion of chemotherapy in that setting.
* Inadequate laboratory parameters defined by:
* Absolute neutrophil count (ANC) < 1,500/μl (1.5x109/L).
* Platelets < 100,000/μl (100x109/L).
* Haemoglobin < 9.0 g/dl or requiring transfusions.
* Creatinine clearance < 45 ml/min (by local institutional methods).
* Total bilirubin outside normal limits:
* ALT and/or AST > 1.5 x ULN in patients without liver metastasis.
* ALT and/or AST > 2.5 x ULN in patients with liver metastasis.
* International normalised ratio (INR) > 2, prothrombin time (PT) and partial thromboplastin time (PTT) > 50% of deviation of institutional ULN.
* Proteinuria CTCAE grade 2 or greater.
* Pre-existing peripheral sensory neuropathy CTCAE grade 2 or greater.
* Use of any investigational drug within 4 weeks of randomisation.
* Radiotherapy within 4 weeks prior to randomisation.
* Major surgery (other than biopsy) within 4 weeks prior to randomisation.
* Active brain metastases or leptomeningeal disease (defined as stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least 4 weeks prior to randomisation).
* Any other active current malignancy (other than non-melanomatous skin cancer, in situ breast or in situ cervical cancer, prostate cancer diagnosed more than 3 years prior, or breast cancer diagnosed more than 5 year prior to randomisation).
* Active or uncontrolled infections or serious illnesses or medical conditions that in the opinion of the investigator could interfere with the patient's participation in the study, including:
* Known active or chronic hepatitis C and/or B infection.
* Known pre-existing interstitial lung disease or pneumonitis
* Presence of significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion).
* Gastro-intestinal abnormalities, including inability to take oral medication, requirement for intravenous feeding, active peptic ulcer, prior surgical procedures affecting absorption, any medical co-morbidity affecting gastrointestinal absorption.
* History of clinically significant haemorrhagic or thromboembolic event in the past 6 months.
* Known inherited predisposition to bleeding or thrombosis.
* Major injuries within the past 10 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
* Drug or alcohol abuse.
* Therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of indwelling intravenous device) or anti-platelet therapy (except low dose therapy with acetylsalicylic acid <325mg her day).
* Radiographic evidence (CT or MRI) of cavitary or necrotic tumours or local invasion of major blood vessels by tumour.
* Pregnancy or breast feeding; female patients must have a negative pregnancy test (beta-HCG test in urine or serum) prior to commencing study treatment.
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception during the trial and for at least three months after ceasing study therapy (medically acceptable methods of contraception include total true abstinence*, permanent sterilisation (see section 7.1.4), combined oral, transdermal or intra-vaginal hormonal contraceptives, methoxyprogesterone injections (e.g. Depo-provera), copper-banded intra-uterine devices, hormone-impregnated intra-uterine systems and vasectomised partners; all methods of contraception, with the exception of total abstinence, should be used in combination with the use of a condom by male sexual partners).
* Known hypersensitivity or any contraindications to the trial drugs, including nab-paclitaxel/nintedanib, to their excipients or to contrast media or other ingredients including peanuts and soya.
* Patients unable to comply with the protocol.

  * True abstinence, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to IMP, and withdrawal are not acceptable methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum Tolerated Dose | 1 and 2 years from patients commencement
  To define Maximum tolerated dose (MTD) and evaluate incidence of dose-limiting toxicities (DLTs) during Cycle 1

SECONDARY OUTCOMES:
Part 1 and 2: Adverse Events Review | 4 years from Start date of trial
  To examine the frequency of all Adverse Events graded by NCI-CTCAE version 4.0
Part 1 and 2: RECIST Response | 4 years from start date of trial
  To examine the objective tumour response according to RECIST 1.1
Cycles Tolerated | 4 years from start date of trial
  To define the number of cycles of nab-paclitaxel with nintedanib given
Part 2: Overall Survival | 9 months post Chemotherapy
  To examine overall survival in the ITT and predefined subgroups (PD pre/post 9 months from start of first line chemotherapy; prior or no prior immunotherapy).

OTHER OUTCOMES:
Part 2: Progression Free Survival | 12 weeks post first dose of treatment and ongoing until end of study
  To explore PFS rate at 12 weeks from first dose of nab-paclitaxel with nintedanib/placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Popat, Principal Investigator — Royal Marsden NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No